CLINICAL TRIAL: NCT05154643
Title: Quantitative Rotating Frame Relaxometry for Early Detection of Liver Fibrosis in Presence of Hepatic Iron
Brief Title: T1rho Imaging of Liver in Presence of Iron
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Weitian, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2018.235
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Liver Fibrosis
Keywords: Quantitative rotating frame relaxometry, T1rho, early detection of liver fibrosis, hepatic iron
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with liver fibrosis
- healthy controls

SUMMARY:
Liver T1rho is elevated in response to accumulation of extracellular matrix proteins during fibrosis. The presence of hepatic iron overload; however, can shorten the T1rho value. With proper correction, we can remove this confounding factor and improve the reliability of T1rho for early diagnosis of liver fibrosis.

Patients with early-stage liver fibrosis confirmed by biopsy will be recruited at the Prince of Wales Hospital (Hong Kong). Thirty patients and twenty healthy volunteers will be recruited. The liver iron content will be measured using the established T2* MRI relaxometry. Breathhold black blood T1rho relaxometry will be used to collect T1rho data. The measured T1rho will be retrospectively corrected to remove the shortening effect caused by iron.

We will use ANOVA to compare the measurement with and without fibrosis. We will use Pearson correlations between the disease state and the imaging measurements, and ROC analysis to determine the diagnostic value of the proposed method.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18 and age 55
* Informed written consent obtained

Exclusion Criteria:

* Contraindications to MRI such as the presence of metallic implants, claustrophobia and pregnancy

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patients with liver fibrosis and healthy controls will be screened before receiving MR exam.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The liver iron content will be measured using the established T2* MRI relaxometry | one year
  Breathhold black blood T1rho relaxometry will be used to collect T1rho data. The measured T1rho will be retrospectively corrected to remove the shortening effect caused by iron.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong